CLINICAL TRIAL: NCT03910608
Title: The Mechanisms of Cortico-cortical and Cortico-subcortical Networks in Methamphetamine Addiction by Paired Associative Stimulation
Brief Title: Paired Associative Stimulation in Methamphetamine Addiction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Haifeng Jiang, associate chief physician, Shanghai Mental Health Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: HFJiang-003
Record Dates: First submitted 2019-04-05; First posted 2019-04-10 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Methamphetamine-dependence
Keywords: Paired Associative Stimulation; Frontoparietal Pathway; Transcranial Magnetic Stimulation; Cognitive Function

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- DLPFC+10 IPL (Experimental): Stimulation of dorsolateral prefrontal cortex (DLPFC) 10 ms before inferior parietal lobule (IPL) presumes that the DLPFC to IPL input facilitates insula postsynaptic output activity, thereby improving cognition response via a long term potentiation-like effect.
  Interventions: Device: MagPro X100 device (MagVenture, Farum, Denmark)
- IPL+10 DLPFC (Experimental): Stimulation of IPL 10 ms before DLPFC presumes that the IPL to DLPFC input inhibits insula postsynaptic output activity, thereby impairing cognition response via a long term depression-like effect.
  Interventions: Device: MagPro X100 device (MagVenture, Farum, Denmark)
- IPL+4 DPLFC (Experimental): Stimulation of IPL 4 ms before DLPFC is presumed to be too brief for a corticocortical effect but presumes that the DLPFC input to insula inhibits insula postsynaptic output by weakening the IPL to insula input, thereby impairing cognition response.
  Interventions: Device: MagPro X100 device (MagVenture, Farum, Denmark)
- DLPFC+4 IPL (Experimental): Stimulation of DLPFC 4 ms before IPL is presumed to be too brief for a corticocortical effect but presumes that the DLPFC input to insula potentiates insula postsynaptic output by strengthening the IPL to insula input, thereby improving cognition response.
  Interventions: Device: MagPro X100 device (MagVenture, Farum, Denmark)
- DLPFC+4 MPFC (Experimental): Stimulation of DLPFC 4 ms before medial prefrontal cortex (MPFC) presumes that the DLPFC input facilitates MPFC postsynaptic output activity, thereby improving cognition response via a long term potentiation-like effect.
  Interventions: Device: MagPro X100 device (MagVenture, Farum, Denmark)
- MPFC+4 DLPFC (Experimental): Stimulation of MPFC 4 ms before DLPFC presumes that the DLPFC input inhibits MPFC postsynaptic output activity, thereby impairing cognition response via a long term depression-like effect.
  Interventions: Device: MagPro X100 device (MagVenture, Farum, Denmark)
- DLPFC+10 MPFC (Experimental): Stimulation of DLPFC 10 ms before medial prefrontal cortex (MPFC) presumes that the DLPFC input facilitates MPFC postsynaptic output activity, thereby improving cognition response via a long term potentiation-like effect.
  Interventions: Device: MagPro X100 device (MagVenture, Farum, Denmark)
- MPFC+10 DLPFC (Experimental): Stimulation of MPFC 10 ms before DLPFC presumes that the DLPFC input inhibits MPFC postsynaptic output activity, thereby impairing cognition response via a long term depression-like effect.
  Interventions: Device: MagPro X100 device (MagVenture, Farum, Denmark)

INTERVENTIONS:
Device: MagPro X100 device (MagVenture, Farum, Denmark) — Each cPAS experimental session contained 100 pairs of stimuli at 0.2 Hz. The experimental conditions differed in the interstimulus interval of the paired pulses. DLPFC stimulation precedes IPL/MPFC stimulation by 10 ms (DLPFC+10) or by 4 ms (DLPFC+4), and IPL/MPFC stimulation precedes DLPFC stimulation by 4 ms (IPL/MPFC+4) or by 10 ms (IPL+10).

SUMMARY:
The investigators use paired associative stimulation (PAS) protocols to target cortico-cortical and cortico-subcortical networks to study cognitive deficits in methamphetamine addiction.

DETAILED DESCRIPTION:
Paired associative stimulation (PAS) is a form of transcranial magnetic stimulation in which paired pulses can induce plasticity at cortical synapses, producing long-term potentiation (LTP) or long-term depression (LTD) effect. The investigators use paired associative stimulation (PAS) protocols to target cortico-cortical and cortico-subcortical networks (frontoparietal control pathway) by using different intervals between the paired pulses to explore the mechanism of cognitive deficits in methamphetamine addiction. The investigators hypothesize that different temporal sequences of cortical stimulation could produce facilitation or inhibition effect.

ELIGIBILITY:
Inclusion Criteria:

* In accordance with the Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) for methamphetamine (MA) use disorders
* Junior high school degree or above
* Normal vision and hearing
* Dextromanual

Exclusion Criteria:

* Have a disease that affect cognitive function such as history of head injury, cerebrovascular disease, epilepsy, etc
* Have cognitive-promoting drugs in the last 6 months
* Other substance abuse or dependence in recent five years (except nicotine)
* Mental impairment, Intelligence Quotient (IQ) < 70
* Mental disorders
* Physical disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Change of working memory | 30 minutes
  The N-Back is a working memory task where the subject is presented with a sequence of stimuli (letters). The task consists of indicating when the current stimulus matches the one from n steps earlier in the sequence.
Change of response inhibition | 30 minutes
  Response inhibition was assessed with the SST (Cambridge Cognition, Cambridge, UK). The subject responded to an arrow (go signal), pointing either right or left, by pressing one of two buttons with the right or left index finger. If an audio tone (stop signal) was present, the subject needed to withhold the response.
Change of attention bias | 30 minutes
  During the dot-probe task, participants are situated in front of a computer screen with their chin securely placed on a chin rest. Participants are asked to stare at a fixation cross on the center of the screen. Two stimuli, one of which is neutral and one of which is threatening, appear randomly on either side of the screen. The stimuli are presented for a predetermined length of time (most commonly 500ms), before a dot is presented in the location of one former stimulus. Participants are instructed to indicate the location of this dot as quickly as possible, either via keyboard or response box.
Change of risk decision | 30 minutes
  The Balloon Analogue Risk Task (BART) is a computerized measure of risk taking behavior. In the task, the participant is presented with a balloon and offered the chance to earn money by pumping the balloon up by clicking a button. Each click causes the balloon to incrementally inflate and money to be added to a counter up until some threshold, at which point the balloon is over inflated and explodes.

SECONDARY OUTCOMES:
Change of eeg oscillatory (Alpha, Beta, Theta and Delta) | 30 minutes
  EEG was recorded to evaluate the changes in the oscillatory domain before and after the stimulation.
Change of eeg functional connectivity (Alpha, Beta, Theta and Delta) | 30 minutes
  EEG was recorded to evaluate the changes of functional connectivity before and after the stimulation.
Change of motor evoked potential | 30 minutes
  Single-pulse TMS will be used to evoke a motor response that is recorded using electromyography (EMG). The peak-to-peak amplitude of the EMG response will be measured.
Change of resting motor threshold | 30 minutes
  Single-pulse TMS will be used to evoke a motor response that is recorded using electromyography (EMG). The lowest stimulator output needed to elicit a consistent response will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Haifeng Jiang, PhD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Haifeng Jiang, Shanghai, Shanghai Municipality, China